CLINICAL TRIAL: NCT02813265
Title: A Phase 3, Double-Masked, Randomized, Controlled Study of KPI-121 0.25% Ophthalmic Suspension Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: Safety and Efficacy of KPI-121 in Subjects With Dry Eye Disease
Acronym: STRIDE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kala Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPI-121-C-006
Record Dates: First submitted 2016-06-21; First posted 2016-06-24 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Dry Eye Syndromes; Keratoconjunctivitis Sicca
Keywords: Ocular Discomfort; Pain; Corticosteroid; Hyperemia; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca; Pain; Hyperemia | interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KPI-121 0.25% Ophthalmic Suspension (Active Comparator)
  Interventions: Drug: KPI-121 0.25% Ophthalmic Suspension
- Vehicle of KPI-121 0.25% Ophthalmic Suspension (Placebo Comparator)
  Interventions: Drug: Vehicle of KPI-121 0.25% Ophthalmic Suspension

INTERVENTIONS:
Drug: KPI-121 0.25% Ophthalmic Suspension
  Other Names: Loteprednol etabonate
  Arms: KPI-121 0.25% Ophthalmic Suspension
Drug: Vehicle of KPI-121 0.25% Ophthalmic Suspension
  Other Names: Placebo
  Arms: Vehicle of KPI-121 0.25% Ophthalmic Suspension

SUMMARY:
The primary purpose of this study is to determine the efficacy and safety of KPI-121 0.25% ophthalmic suspension compared to vehicle (placebo) in subjects who have a documented clinical diagnosis of dry eye disease. The product will be studied over 14 days, with 1-2 drops instilled in each eye four times daily (QID).

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, double-masked, randomized, vehicle-controlled, parallel-group study designed to evaluate the safety and efficacy of KPI-121 0.25% ophthalmic suspension versus vehicle in subjects with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented clinical diagnosis of dry eye disease in both eyes

Exclusion Criteria:

* Known hypersensitivity or contraindication to the investigational product(s) or components
* History of glaucoma, Intraocular Pressure (IOP) >21 mmHg at the screening or randomization visits, or being treated for glaucoma in either eye.
* Diagnosis of: ongoing ocular infection; severe/serious ocular condition that in judgment of Investigator could confound study assessments or limit compliance; or have been exposed to an investigational drug within 30 days prior to screening.
* In the opinion of the Investigator or study coordinator, be unwilling or unable to comply with study protocol or unable to successfully instill eye drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 918 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (60):
  - Cornea and Cataract Consultants of Arizona, Phoenix, Arizona
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - Eyecare Arkansas, P.A., Little Rock, Arkansas
  - Little Rock Eye Clinic, LLP, Little Rock, Arkansas
  - Sall Research Medical Center, Artesia, California
  - Orange County Ophthalmology Medical Group, Garden Grove, California
  - United Medical Research Institute, Inglewood, California
  - North Valley Eye Medical Group, Mission Hills, California
  - Montebello Medical Center, Inc., Montebello, California
  - LoBue Laser and Eye Medical Center, Murrieta, California
  - Eye Research Foundation, Newport Beach, California
  - Pendleton Eye Center, Oceanside, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Sacramento Eye Consultants, Sacramento, California
  - Eye Center of Northern Colorado, PC, Fort Collins, Colorado
  - Corneal Consultants of Colorado, Littleton, Colorado
  - The Eye Center of Southern CT, P.C., Hamden, Connecticut
  - Florida Eye Microsurgical Institute, Inc., Boynton Beach, Florida
  - Eye Associates of Fort Myers, Fort Myers, Florida
  - Shettle Eye Research, Inc., Largo, Florida
  - Atlantic Eye Center, Palm Coast, Florida
  - The Eye Center of North Florida, Panama City, Florida
  - Dixon Eye Care, Albany, Georgia
  - Jacksoneye, S. C., Lake Villa, Illinois
  - Midwest Cornea Associates, LLC, Indianapolis, Indiana
  - Stiles EyeCare Excellence and Glaucoma Institute, Overland Park, Kansas
  - Clinical Eye Research of Boston, Winchester, Massachusetts
  - Chu Vision Institute, Bloomington, Minnesota
  - Lifelong Vision Foundation at Pepose Vision Institute, Chesterfield, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Ophthalmology Consultants, Ltd., St Louis, Missouri
  - Wellish Vision Institute, Las Vegas, Nevada
  - Matossian Eye Associates, Pennington, New Jersey
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - Cornea Consultants of Albany, Slingerlands, New York
  - South Shore Eye Center, LLP, Wantagh, New York
  - Mundorf Eye Center, Charlotte, North Carolina
  - Firozvi Research, LLC / North Carolina Eye, Ear, Nose & Throat, Durham, North Carolina
  - Eyecare Center, Raleigh, North Carolina
  - Bergstrom Eye Research, Fargo, North Dakota
  - Abrams Eye Center, Cleveland, Ohio
  - Opthalamic Surgeons & Consultants of Ohio, Columbus, Ohio
  - Apex Eye, Mason, Ohio
  - Roseburg Research Associates, LLC, Roseburg, Oregon
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Conestoga Eye, Lancaster, Pennsylvania
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Total Eye Care, PA, Memphis, Tennessee
  - Hill Country Eye Center, Cedar Park, Texas
  - Houston Eye Associates, Houston, Texas
  - The Eye Clinic of Texas, Affiliate of Houston Eye Associates, League City, Texas
  - Lake Travis Eye and Laser Center, Leander, Texas
  - Eye Clinics of South Texas, San Antonio, Texas
  - R and R Eye Research, LLC, San Antonio, Texas
  - Keystone Research - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Tanner Clinic, Layton, Utah
  - See Clearly Vision, McLean, Virginia
  - Virginia Eye Consultants, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 918 subjects were randomized, 3 of which were not included in any analysis population as they had participated in more than one study. The data for the second-participation for these 3 individuals were not included in any analysis population as agreed upon with the FDA.
Groups:
- KPI-121 0.25% Ophthalmic Suspension: Participants randomized to KPI-121 0.25% Ophthalmic Suspension
- Vehicle of KPI-121 0.25% Ophthalmic Suspension: Participants randomized to Vehicle of KPI-121 0.25% Ophthalmic Suspension
Period: Overall Study
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Started | 459 | 456
Completed | 455 | 453
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension | Total
Number analyzed (Participants) | 459 | 456 | 915
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (15.41) | 58.3 (14.66) | 58.2 (15.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 367 | 359 | 726
  Male | 92 | 97 | 189
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 18 | 18 | 36
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 69 | 71 | 140
  White | 362 | 361 | 723
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 459 | 456 | 915

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline/Visit 2 (Day 1) in Bulbar Conjunctival Hyperemia at Visit 4 (Day 15)
Description: Comparison of mean bulbar conjunctival hyperemia between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-4 grading scale. The grading scale was based on the Cornea and Contact Lens Research Unit Grading Scale where 0 = none, 1 = very slight, 2 = slight, 3 = moderate and 4 = severe.
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 4 (Day 15)
Population: Intent to Treat population minus subjects in each treatment group that discontinued the study by this time point or otherwise did not have this assessment completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 452 | 451
score on a scale | -0.4049 (0.65062) | -0.1574 (0.60704)

2. Primary Outcome: Change From Baseline/Visit 2 (Day 1) in Ocular Discomfort Severity at Visit 4 (Day 15)
Description: Comparison of mean ocular discomfort severity between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-100 visual analog grading scale where 0 was better and 100 was worse.
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 4 (Day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 455 | 452
score on a scale | -14.53 (20.636) | -9.16 (17.924)

3. Primary Outcome: Change From Baseline/Visit 2 (Day 1) in Corneal Fluorescein Staining Score at Visit 4 (Day 15)
Description: Comparison of mean corneal fluorescein staining between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using methods developed by the National Eye Institute (NEI) Dry Eye Workshop in evaluating 5 regions of the cornea (superior, inferior, nasal, temporal and central) using a 0-3 grading scale, where 0 = no visible staining, 1 = Mild, 2 = moderate and 3 = severe.
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 4 (Day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 455 | 452
score on a scale | -0.5 (0.84) | -0.4 (0.79)

4. Primary Outcome: Change From Baseline/Visit 2 (Day 1) Ocular Discomfort Severity at Visit 4 (Day 15) in the Subgroup of Participants With More Severe Ocular Discomfort
Description: Comparison of mean ocular discomfort severity between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-100 visual analog grading scale where 0 was better and 100 was worse, in a sub-group of participants with more severe ocular discomfort at baseline.
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 4 (Day 15)
Population: Sub-group of Intent to Treat population with more severe ocular discomfort minus subjects in each treatment group that discontinued the study by this time point or otherwise did not have this assessment completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 233 | 238
score on a scale | -16.67 (21.937) | -10.76 (18.037)

5. Secondary Outcome: Change in Conjunctival Hyperemia Scores at Visit 4 (Day 15) in the Subgroup of Participants With More Severe Ocular Discomfort at Baseline (Day 1)
Description: as for outcome 1
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 4 (Day 15)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 256 | 264
score on a scale | -0.4648 (0.66770) | -0.2045 (0.62567)

6. Secondary Outcome: Proportion of Subjects With ≥1 Improvement in Conjunctival Hyperemia at Visit 4 (Day 15)
Description: Proportion of subjects with ≥1 improvement from baseline in conjunctival hyperemia scores. The grading scale was based on the Cornea and Contact Lens Research Unit Grading Scale where 0 = none, 1 = very slight, 2 = slight, 3 = moderate and 4 = severe.
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 4 (Day 15)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 452 | 451
Participants | 189 | 98

7. Secondary Outcome: Change From Baseline/Visit 2 (Day 1) Conjunctival Hyperemia Scores at Visit 4 (Day 15) for the Mean of All Regions (Nasal, Temporal, Frontal)
Description: as for outcome 1
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 4 (Day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 453 | 450
score on a scale | -0.2980 (0.59018) | -0.0421 (0.51921)

8. Secondary Outcome: Change in Ocular Discomfort Severity Scores Prior to Visit 3 (Day 8) Minus the Mean of the Scores to Baseline/Visit 2 (Day 1)
Description: as for outcome 2
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 3 (Day 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 457 | 455
score on a scale | -8.12 (16.880) | -4.81 (14.851)

9. Secondary Outcome: Change in Ocular Discomfort Severity Scores Prior to Visit 3 (Day 8) Minus Baseline/Visit 2 (Day 1) in the Subgroup of Participants With More Severe Ocular Discomfort.
Description: as for outcome 2
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 3 (Day 8)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 258 | 263
score on a scale | -9.90 (17.835) | -6.38 (15.289)

10. Secondary Outcome: Change in Ocular Discomfort Severity Scores on Day 4 (Diary) Minus Baseline/Visit 2 (Day 1)
Description: as for outcome 2
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 3 (Day 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 455 | 452
score on a scale | -6.60 (16.710) | -3.20 (15.125)

11. Secondary Outcome: Change in Ocular Discomfort Severity Scores on Day 4 Day 4 (Diary) Minus Baseline/Visit 2 (Day 1) in the Subgroup of Participants With More Severe Ocular Discomfort
Description: as for outcome 4
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 3 (Day 8)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 256 | 261
score on a scale | -8.48 (17.412) | -5.20 (14.903)

12. Secondary Outcome: Change From Baseline/Visit 2 (Day 1) in Conjunctival Hyperemia Scores With a Day 1 Conjunctival Hyperemia Score of ≥ 2 in the Subgroup of Participants With More Severe Ocular Discomfort
Description: Comparison of mean bulbar conjunctival hyperemia between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-4 grading scale in a sub-group of participants with more severe ocular discomfort at baseline.. The grading scale was based on the Cornea and Contact Lens Research Unit Grading Scale where 0 = none, 1 = very slight, 2 = slight, 3 = moderate and 4 = severe.
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 4 (Day 15)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 379 | 379
score on a scale | -0.47 (0.631) | -0.22 (0.577)

13. Secondary Outcome: Subjects With a Grade of 0 in Conjunctival Hyperemia Score at Visit 4 (Day 15)
Description: as for outcome 1
Time Frame: Visit 4 (Day 15)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 453 | 451
Participants | 27 | 16

ADVERSE EVENTS:
Time Frame: Adverse events were collected at Visit 2 (Day 1) until they exited the study at Visit 4 (Day 15).
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
All-Cause Mortality (participants affected / at risk) | 0/459 | 0/456
Serious Adverse Events (participants affected / at risk) | 0/459 | 0/456
Other Adverse Events (participants affected / at risk) | 66/459 | 62/456
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KPI-121 0.25% Ophthalmic Suspension (N=459) | Vehicle of KPI-121 0.25% Ophthalmic Suspension (N=456)
Eye Irritation (Eye disorders) | 5 | 7
Blepharitis (Eye disorders) | 3 | 0
Lacrimination increased (Eye disorders) | 3 | 2
Conjunctival hyperemia (Eye disorders) | 2 | 4
Eye Pain (Eye disorders) | 2 | 1
Foreign Body Sensation (Eye disorders) | 2 | 4
Conjunctival vascular disorder (Eye disorders) | 1 | 0
Eye discharge (Eye disorders) | 1 | 0
Eye Pruritus (Eye disorders) | 1 | 4
Eyelid margin crusting (Eye disorders) | 1 | 2
Eyelid ptosis (Eye disorders) | 1 | 0
Trichiasis (Eye disorders) | 1 | 0
Vision Blurred (Eye disorders) | 1 | 2
Vitreous detachment (Eye disorders) | 1 | 0
Blepharospasm (Eye disorders) | 0 | 1
Keratitis (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 1
Punctate keratitis (Eye disorders) | 0 | 1
hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Installation site pain (General disorders) | 28 | 28
Instillation site foreign body sensation (General disorders) | 2 | 0
Instillation site lacrimation (General disorders) | 1 | 0
Instillation site pruritus (General disorders) | 1 | 3
Installation site discomfort (General disorders) | 0 | 1
Installation site reaction (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Intraocular pressure increased (Investigations) | 3 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Nerve Compression (Nervous system disorders) | 1 | 0
Sinus Headache (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0
Eccymosis (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement between the Principal Investigator and the Sponsor restricts the PI's rights to discuss or publish trial results until after the first to occur of the following:

(a) publication of such multi-center clinical trial results; (b) notification by sponsor that such a multi-center clinical trial submission is no longer planned; or ( c) the eighteen ( 18) month anniversary of the completion, abandonment or termination of such multi-center clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT02813265/Prot_SAP_000.pdf